CLINICAL TRIAL: NCT06583278
Title: The Efficacy of Repetitive Transcranial Magnetic Stimulation in Parkinson's Disease：A Randomized, Double-blind, Multicenter, Placebo-controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Head, Dept of Neurology & Medical Psychology, Director, Cognitive Neuropsychology Lab, PRC, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHMU-PPD
Record Dates: First submitted 2024-09-01; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease; Transcranial Magenetic Stimualtion; Supplementary Motor Area
Keywords: Parkinson Disease; Transcranial Magenetic Stimualtion; Supplementary Motor Area
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real rTMS group (Active Comparator): Participants will receive real transcranial magnetic stimulation (TMS) daily for 1 week.
  Interventions: Device: transcranial magnetic stimulation
- Sham rTMS group (Sham Comparator): Participants will receive sham transcranial magnetic stimulation (TMS) daily for 1 week.
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — The stimulations were performed by MagStim Rapid2.

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive and widely used neuromodulation technology. Small sample studies have shown that rTMS treatment can significantly improve the symptoms of Parkinson's disease(PD) and delay the progression of the disease. In order to further explore the effectiveness of rTMS in the treatment of PD and lay the foundation for its clinical promotion, our research team plans to conduct a randomized double-blind controlled study of rTMS in the treatment of PD in multiple centers across the country.

DETAILED DESCRIPTION:
As an innovative non-invasive neuromodulation technology, repetitive transcranial magnetic stimulation (rTMS) has demonstrated efficacy in improving motor symptoms in patients with Parkinson's disease (PD). The supplementary motor area (SMA) has been identified as a brain region significantly associated with motor symptoms in PD patients. However, no large-sample clinical studies have yet established the clinical efficacy of rTMS, guided by neuroimaging navigation, targeting the SMA in patients with Parkinson's disease.

We describe a randomized, controlled, double-blind, placebo-treated, multicenter study designed to recruit 312 patients with idiopathic Parkinson's disease. Participants will be randomly assigned to receive either real stimulation or sham stimulation, with the left SMA undergoing 7 days of continuous theta burst stimulation (cTBS). The primary outcome measure is the change in the Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III scores from baseline to post-treatment and follow-up. Secondary outcomes include changes in scores on other clinical symptom scales. The study is expected to be conducted across nine medical centers in China, commencing in 2024 and concluding in 2026.

This study will evaluate the clinical efficacy of cTBS targeting the left SMA in patients with Parkinson's disease. The findings may offer a new therapeutic approach for PD.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥40 years old
2. Meet Movement Disorder Society standards;
3. Have no history of drug adjustment within 4 weeks before and during treatment;
4. The MDS-UPDRS Ⅲ score ≥8, and the Hoehn-Yahr rating is 1-4
5. MMSE ≥24，able to cooperate with the completion of behavioral tests and transcranial magnetic stimulation therapy.

Exclusion Criteria:

1. Head MRI/CT ruled out focal brain injury or severe leukoencephalopathy (Fazekas grade 3);
2. Various secondary parkinsonism syndromes (vascular parkinsonism, Parkinsonism combined with parkinsonism, drug parkinsonism, etc.);
3. Severe craniocerebral trauma, received craniocerebral surgery or deep brain stimulation treatment;
4. There are ferromagnetic implants in the body, such as cochlear implants, cardiac pacemakers, etc.
5. The person or first-degree relatives have a history of epilepsy, unexplained loss of consciousness, or are taking anticonvulsant drugs to treat epileptic seizures;
6. Diagnosed with a neuropsychiatric disorder other than PD
7. Have a history of drug abuse or drug use;
8. Participants in any clinical trial within the previous 6 month;
9. Pregnant/lactating women or subjects (including men) who have a birth plan within 6 months;
10. Other conditions deemed unsuitable for inclusion by the investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society- Unified Parkinson's Disease Rating Scale III scores | baseline; day 8; week 5;week 9
  This is an very common clinical motor estimating scale with 18 items and 140' in total. Higher scores indicate worse symptoms.

SECONDARY OUTCOMES:
Movement Disorder Society- Unified Parkinson's Disease Rating Scale I scores | baseline; day 8; week 5;week 9
  MDS-UPDRS Ⅰ was used to evaluate the experience of non-motor symptoms of daily living in patients with Parkinson's disease. Items 1.1 to 1.6 were asked and evaluated by the raters, including some cognitive impairment, anxiety and depression symptoms, and dopamine dysregulation symptoms. Items 1.7-1.13 were scored by the patients themselves, and the problems involved included sleep, fatigue, urination, constipation, etc.
Movement Disorder Society- Unified Parkinson's Disease Rating Scale Ⅱ scores | baseline; day 8; week 5;week 9
  MDS-UPDRS II is used to evaluate the patient's experience of motor symptoms of daily living, such as speech function, eating capacity, daily living capacity (eating, dressing, hygiene), tremor, walking, etc.
Movement Disorder Society- Unified Parkinson's Disease Rating Scale Ⅳ scores | baseline; day 8; week 5;week 9
  The MDS-UPDRS Ⅳ questionnaire consisted of raters combining previously known and objective information on patients with two motor complications: motor fluctuations and AIMs. All three segments are rated on a 0-4 scale.
Hoehn-Yahr(H-Y) scale | baseline; day 8; week 5;week 9
  H-Y scale is a standardized instrument used to evaluate the severity of Parkinson's disease. It employs a scoring system that ranges from 1 to 5, with higher scores indicating greater severity of clinical symptoms and a corresponding decline in quality of life. The assessment criteria primarily consider the number of limbs affected, the presence of balance disturbances, and the extent of functional impairment in daily living activities. This scale is valued for its simplicity and practicality, making it a prevalent tool in clinical trials for evaluating Parkinson's disease symptoms.
The timed up and go test (TUG) | baseline; day 8; week 5;week 9
  TUG measures in seconds how long it takes the subject to rise from the chair, walk 3 meters, turn around, walk back to the chair, and sit down. The test is often used to assess walking and balance in older adults. This also applies to evaluating the severity of walking and balance symptoms in patients with Parkinson's disease.
20 meters walking | baseline; day 8; week 5;week 9
  The 20-meter walking test measured the time it took for the subject to turn, continue to walk to the original place and turn back after walking from the upright position for 10m in seconds, and recorded the total number of steps. The test is also used to assess walking and balance in people with Parkinson's disease, but the distance is longer and more stable. Both tests were recorded on video with the patient's consent.
Upper and lower limb rotation counting | baseline; day 8; week 5;week 9
  The upper and lower limb alternation count is used to record the total number of times a subject presses or steps on the counter (including both the left and right sides) within a specified 30-second interval. This test assesses the motor function of patients with Parkinson's disease. By observing the changes in the total count before and after treatment, the test evaluates whether the patient's symptoms of bradykinesia have improved.
Non-motor symptom scale（NMSS） | baseline; day 8; week 5;week 9
  NMSS is a validated assessment tool for non-motor symptoms in patients with PD. The scale consists of nine domains, each carrying a separate domain score, with higher scores indicating more severe symptoms for that domain. The score for each domain is derived by multiplying the severity and frequency ratings on a scale of 0-4. The total NMSS score is the sum of the nine field scores.
Clinical Global Impression（CGI） | baseline; day 8; week 5;week 9
  CGI is used to evaluate the clinical treatment effect and is conducted by uniformly trained evaluators. The scale consists of three parts: severity of illness (SI), global improvement (GI) and efficacy index (EI). When evaluating SI, it is necessary to evaluate the severity of the patient's disease according to the relevant experience of patients with the same diagnosis in the past. When evaluating GI, the evaluator should compare the current condition of the patient with that at the time of enrollment to evaluate the treatment effect of the patient. Both SI and GI are evaluated on a scale of 0-7. Evaluation of EI includes two aspects, namely efficacy and side effects caused by treatment. Both were rated on a scale of 1-4. EI= efficacy score/side effect score. This scale integrates the severity of the patient's disease and the effect of treatment, which is helpful for following up the patient's condition changes.
Parkinson's Disease questionnaire-39 items（PDQ-39） | baseline; day 8; week 5;week 9
  PDQ-39 is a self-rating scale for clinical evaluation of the quality of life of patients with Parkinson's disease, which consists of 8 dimensions and 39 items. The rating ranges from 0 to 4. The PDQ-39 total score is the sum of the 39 project scores.
Hamilton Depression Scale-17（HAMD-17） | baseline; day 8; week 5;week 9
  HAMD-17 is commonly used in clinical trials to assess the severity of depression and is the gold standard for diagnosing depression. The scale was used to assess the depressive symptoms of patients through conversation and observation by uniformly trained evaluators, including 17 items, scoring on a 0-4 scale. If the total score is <7, there is no depression; A score between 7 and 17 indicates mild depression. A score between 18 and 24 indicates moderate depression; If the total score is more than 24, it indicates major depression.
Hamilton Anxiety Scale（HAMA） | baseline; day 8; week 5;week 9
  HAMA is a tool commonly used to diagnose anxiety disorders. The evaluators with standardized training evaluated the anxiety symptoms of the patients by way of conversation and observation, which were mainly divided into physical anxiety and mental anxiety, with a total of 14 sub-items, the score range was 0-4, and the sum of the scores of each sub-item was the total score of the scale. If the total score is more than 29, it may be severe anxiety; Over 21 points, there must be significant anxiety; If more than 14 points, definitely have anxiety; More than 7 points, may have anxiety; Less than 7, no anxiety.
Pittsburgh sleep quality index（PSQI） | baseline; day 8; week 5;week 9
  PSQI was used to evaluate the sleep quality of patients with sleep disorders and general people in the past month. The scale consists of 4 fill-in-the-blank questions and 5 multiple choice questions, and the fifth multiple choice question includes 10 multiple choice questions, for a total of 18 questions. The questions assessed patients' sleep quality from seven factors, including: subjective sleep quality, time to fall asleep, sleep duration, habitual sleep efficiency, sleep disorders, hypnotic medications, and daytime function. The total score of the scale is the sum of the 7 factor scores. The total score ranges from 0 to 21, with higher scores indicating poorer sleep quality.
Montreal Cognitive Assessment（MoCA） | baseline; day 8; week 5;week 9
  MoCA is an assessment tool for rapid screening of Mild Cognitive Impairment (MCI) in the areas of attention and concentration, executive function, memory, language, visual structure skills, abstract thinking, and computation and orientation on a scale of 30 points. In addition, according to the education level of the subject, the corresponding points should be given. If the subject has no formal education, add 1 point; If the subject has only primary or secondary education, add 2 points; No extra points are given if the subject has a high school education or above.

IPD SHARING:
Plan to Share IPD: No